CLINICAL TRIAL: NCT07391488
Title: Investigation of the Effects of Lumbopelvic Rhythm on Postural Control, Daily Living Activities, and Quality of Life in Adolescent Individuals With Idiopathic Scoliosis
Brief Title: The Effects of Lumbopelvic Rhythm on Postural Control, Daily Activities, and Quality of Life in Individuals With AIS
Acronym: AIS
Status: Enrolling by invitation | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, CEM SAMUT, Lecturer, Hacettepe University
Other Study IDs: FTREK25/59
Record Dates: First submitted 2026-01-09; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Adolescence Idiopathic Scoliosis
Keywords: ADOLESCENT IDIOPATHIC SCOLIOSIS; LUMBOPELVIC RHYTHM; POSTURAL CONTROL

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants diagnosed with scoliosis who are assessed at a single time point for observational meas: Adolescent idiopathic scoliosis 10-18 age

SUMMARY:
Adolescent idiopathic scoliosis (AIS) leads to three-dimensional spinal deformity during adolescence, causing deviations in the frontal, sagittal, and axial planes, impairing physical function, balance, and lumbopelvic rhythm. Individuals with AIS exhibit decreased trunk movement, muscle overactivation, increased energy expenditure, balance/gait disturbances, and abnormalities in proprioceptive/vestibular input; pressure center deviations increase in postural control. These changes negatively impact daily life, pain, and quality of life.

Although the literature has examined the relationships between AIS and muscle activation, range of motion, pelvic position, and gait/balance, the relationship between lumbopelvic rhythm changes and curve type/localization/severity, and its impact on postural control and quality of life, has not been investigated. This study aims to elucidate movement patterns by evaluating lumbopelvic rhythm in individuals with AIS and to guide clinical diagnosis/treatment.

DETAILED DESCRIPTION:
Adolescent idiopathic scoliosis (AIS) is a condition that emerges during adolescence and causes a three-dimensional deformity of the spine. This deformity can cause deviations in frontal, sagittal, and axial flight, negatively impacting physical function and balance control mechanisms. Lumbopelvic rhythm ensures the coordination of spinal and pelvic movements and is a critical factor for postural stability. Scoliosis can disrupt lumbopelvic rhythm by affecting pelvic and lumbar region movements. Individuals with AIS have been observed to exhibit changes such as decreased trunk flexion-extension movements and pelvic and hip movements during gait, overactivity of muscles involved in the spine and pelvis, increased energy expenditure, and changes in balance and limb alignment. Abnormalities in vestibular and proprioceptive input have also been observed, leading to changes in balance control. Postural control requires the integration of sensory and motor systems to maintain body balance. In individuals with scoliosis, changes in postural control can reduce mobility. Assessments of postural control, when compared to healthy individuals, have shown that those with scoliosis exhibit higher deviations and acceleration rates in pressure points. This can lead to difficulties in daily living activities, increased pain levels, and decreased quality of life. While the literature examines muscle activation, spinal range of motion, pelvic position, gait, and balance in individuals with AIS, studies on the distribution of lumbopelvic rhythm and its relationship to curvature type, localization, and work, as well as the impact of lumbopelvic rhythm on postural control and quality of life, have not been found. Therefore, evaluating lumbopelvic rhythm in individuals with AIS can contribute to a comprehensive understanding of changes in scoliosis-related movement patterns, guiding clinical diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for the AIS group:
* Individuals diagnosed with AIS,
* Aged between 10-18 years,
* Having a Cobb angle greater than 10°,
* Having a pain intensity < 3,
* Volunteer individuals.

Exclusion Criteria:

* Male gender,
* Body mass index ≥30,
* Presence of additional pathologies affecting the lumbopelvic region (disc herniation, spondylolisthesis, hip dysplasia, rheumatic diseases, etc.),
* Chronic pain lasting longer than 3 months,
* Lower extremity length discrepancy > 2 cm,
* Orthopedic or neurological problems affecting the lower or upper extremity,
* History of acute injury,
* History of spinal surgery,
* Individuals with vestibular pathology or severe balance disorders.

Ages: 10 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Only individuals who identify as female are eligible to participate in this study.
Study Population: The study group will consist of individuals diagnosed with AIS who apply to the Faculty of Physical Therapy and Rehabilitation at Hacettepe University. Participants in the healthy group will be selected using a snowball method from among the relatives of patients who apply to the Faculty of Physical Therapy and Rehabilitation or from among the relatives of the researchers.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-12-30 (Actual); Primary Completion 2026-04-08 (Estimated); Study Completion 2026-10-08 (Estimated)

PRIMARY OUTCOMES:
Lumbopelvic rhythm, | January 30, 2025 - October 8, 2026
  An Inertial Measurement Unit (IMU) will be used to assess lumbopelvic rhythm
Postural control | January 30, 2025 - October 8, 2026
  Postural control will be assessed using the Bertec Balance Check Screener™ strength platform (BP5050 Bertec Co., Columbus, OH, USA) (13).

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Çorum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Piatek E, Kuczynski M, Ostrowska B. Postural control in girls with adolescent idiopathic scoliosis while wearing a Cheneau brace or performing active self-correction: a pilot study. PeerJ. 2019 Aug 29;7:e7513. doi: 10.7717/peerj.7513. eCollection 2019. PMID 31528504
- [Background] Pialasse JP, Descarreaux M, Mercier P, Simoneau M. Sensory reweighting is altered in adolescent patients with scoliosis: Evidence from a neuromechanical model. Gait Posture. 2015 Oct;42(4):558-63. doi: 10.1016/j.gaitpost.2015.08.013. Epub 2015 Sep 6. PMID 26371828
- [Background] Pialasse JP, Descarreaux M, Mercier P, Blouin J, Simoneau M. The Vestibular-Evoked Postural Response of Adolescents with Idiopathic Scoliosis Is Altered. PLoS One. 2015 Nov 18;10(11):e0143124. doi: 10.1371/journal.pone.0143124. eCollection 2015. PMID 26580068
- [Background] Mahaudens P, Thonnard JL, Detrembleur C. Influence of structural pelvic disorders during standing and walking in adolescents with idiopathic scoliosis. Spine J. 2005 Jul-Aug;5(4):427-33. doi: 10.1016/j.spinee.2004.11.014. PMID 15996612
- [Background] Mahaudens P, Raison M, Banse X, Mousny M, Detrembleur C. Effect of long-term orthotic treatment on gait biomechanics in adolescent idiopathic scoliosis. Spine J. 2014 Aug 1;14(8):1510-9. doi: 10.1016/j.spinee.2013.08.050. Epub 2013 Oct 4. PMID 24314903
- [Background] Abdel-Aziem AA, Abdelraouf OR, Ghally SA, Dahlawi HA, Radwan RE. A 10-Week Program of Combined Hippotherapy and Scroth's Exercises Improves Balance and Postural Asymmetries in Adolescence Idiopathic Scoliosis: A Randomized Controlled Study. Children (Basel). 2021 Dec 30;9(1):23. doi: 10.3390/children9010023. PMID 35053648

DOCUMENTS (2):
  • Study Protocol (2026-01-23): https://cdn.clinicaltrials.gov/large-docs/88/NCT07391488/Prot_000.pdf
  • Informed Consent Form (2026-01-23): https://cdn.clinicaltrials.gov/large-docs/88/NCT07391488/ICF_001.pdf